CLINICAL TRIAL: NCT06080204
Title: Real-world Effectiveness of Adjuvant Octreotide Therapy in High Recurrence Risk Patients With Pancreatic Neuroendocrine Tumors
Brief Title: Real-world Study on Adjuvant Octreotide Therapy in pNETs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Guo ShiWei, Clinical Professor, Changhai Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChanghaiH-PP12
Record Dates: First submitted 2023-09-26; First posted 2023-10-12 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-09

CONDITIONS: Pancreatic Neuroendocrine Tumor G2
MeSH Terms: interventions — Octreotide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Octreotide group (Experimental): Patients in the octreotide group received octreotide LAR (Sandostatin® LAR, Novartis Pharmaceuticals Corporation) treatment by deep intramuscular injection at a dose of 30 mg every 28 days for 6-12 months, with the start of clinical intervention following surgery.
  Interventions: Drug: Octreotide LAR
- Control group (No Intervention): No adjuvant therapy after surgery.

INTERVENTIONS:
Drug: Octreotide LAR — Octreotide LAR (Sandostatin® LAR, Novartis Pharmaceuticals Corporation) treatment by deep intramuscular injection at a dose of 30 mg every 28 days for 6-12 months。
  Other Names: Sandostatin
  Arms: Octreotide group

SUMMARY:
Adjuvant therapy in pancreatic neuroendocrine tumors (pNETs) after radical resection lacks evidence-based data and is controversial. Real-world data were clustered to validate whether the long-acting octreotide is a potential candidate for adjuvant therapy in high recurrence risk G2 pNET patients.

DETAILED DESCRIPTION:
Adjuvant therapy for pNETs was proposed as an unmet clinical need by the European Neuroendocrine Tumor Society Group in 2016.1The Clinical Practice Guidelines for pNETs in China recommended initiation of clinical trials to investigate the role of adjuvant therapy for patients with a high-risk of recurrence. To address this unmet clinical need, the investigators initiated this real-world study. The aim of the current study was to assess the impact of octreotide LAR as an adjuvant therapy in reducing recurrence and prolonging survival in Chinese non-metastatic pNETs patients at risk for recurrence.

ELIGIBILITY:
Inclusion Criteria:

* pNETs lesions pathologically classified as WHO grade 2
* Complete surgical resection (R0 or R1 was achieved)
* Adjuvant treatment was performed within 12 weeks after surgery

Exclusion Criteria:

* Stage IV
* Other oncological history
* Previous antineoplastic systemic therapy
* Lack of information/details on recurrence or death.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 411 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Disease-free survival time | From the date of surgery to the date of distant metastasis or recurrence or death due to any cause, whichever came first, assessed up to 120 months
  Disease-free survival time

SECONDARY OUTCOMES:
Overall survival time | From the date of surgery to the date of death due to any cause, whichever came first, assessed up to 120 months
  Overall survival time